CLINICAL TRIAL: NCT02392962
Title: Efectos de la Fatiga en el Rendimiento físico en el Ejercicio de Sentadillas
Brief Title: Dynamic and Static Stretching on Postural Stability, Reaction Time and Countermovement Jump of Sprinters
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Católica San Antonio de Murcia (Other)
Collaborators: University of Jaén (Other)
Responsible Party: Principal Investigator, Natalia Romero-Franco, Asistant Professor, Universidad Católica San Antonio de Murcia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: CEIH 201014-2
Record Dates: First submitted 2015-03-05; First posted 2015-03-19 (Estimated); Last update posted 2015-03-19 (Estimated); Status verified 2015-03

CONDITIONS: Postural Stability
Keywords: proprioception; countermovement jump; postural balance
MeSH Terms: interventions — Muscle Stretching Exercises

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Experimental I (Experimental): This group performed static stretching
  Interventions: Procedure: Static Stretching
- Experimental II (Active Comparator): This group performed dynamic stretching
  Interventions: Procedure: Dynamic Stretching

INTERVENTIONS:
Procedure: Static Stretching — To analyze the immediate effects of static stretching on performance of sprinters
  Arms: Experimental I
Procedure: Dynamic Stretching — To analyze the immediate effects of dynamic stretching on performance of sprinters
  Arms: Experimental II

SUMMARY:
All the athletes should perform a warm-up consisting of five minutes of jogging and static stretching (Experimental Group 1) or dynamic stretching (Experimental Group 2). Before the beginning of the study and right after performing the stretching protocol, the investigators evaluated the unipedal postural stability, the acustic reaction time, the joint position sense of the knee and the countermovement jump of the athletes.

ELIGIBILITY:
Inclusion Criteria:

* National level Sprinters
* Two years or more of experience

Exclusion Criteria:

* Free of injuries in the last six months

Ages: 18 Years to 26 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2014-12; Primary Completion 2014-12 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Change in the unipedal postural balance of athletes | baseline and 15 minutes
  Monopodal postural stability (15 seconds as still as possible on a baropodometric platform in left-leg and right-leg monopodal support)
Change in counter-movement jump of athletes | baseline and 17 minutes
  A maximum vertical jump with counter-movement.
Change in Joint Position Sense of the knee of athletes | baseline and 20 minutes
  Acuity of repositioining a previous position of the knee joint
Change in Acustic Reaction Time of athletes | baseline and 22 minutes
  Time spent to rise the dominant leg after an acustic signal

CONTACTS AND LOCATIONS:
Locations (1):
- University of Jaén, Jaén, Jaén, Spain